CLINICAL TRIAL: NCT00592657
Title: Incidence of Rhabdomyolysis Among Pediatric and Adolescent Patients Admitted for Jimsonweed (Datura Stramonium) Ingestions
Brief Title: Incidence of Rhabdomyolysis Among Patients Admitted With Jimsonweed Ingestions
Status: Completed | Type: Observational
Sponsor: Akron Children's Hospital (Other)
Responsible Party: Martha Blackford PharmD, CHMCA
Other Study IDs: JIMSONWEED
Record Dates: First submitted 2008-01-01; First posted 2008-01-14 (Estimated); Last update posted 2008-07-28 (Estimated); Status verified 2008-07

CONDITIONS: Rhabdomyolysis; Myoglobinuria; Hemoglobinuria
Keywords: retrospective chart review; Jimsonweed ingestion
MeSH Terms: conditions — Rhabdomyolysis; Myoglobinuria; Hemoglobinuria

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Patients diagnosed with rhabdomyolysis and no history of jimsonweed ingestion
- 2: Patients diagnosed with rhabdomyolysis and history of jimsonweed ingestion

SUMMARY:
Retrospective chart review to determine the presence of rhabdomyolysis among patients admitted to CHMCA from 1997-2007 with Jimsonweed ingestions and to define possible risk factors predisposing patients to the developement of Jimsonweed-associated rhabdomyolysis.

ELIGIBILITY:
Inclusion Criteria:

* admitted to CHMCA between 1/1/1997 to 12/31/2007 with a qualifying ICD-9 diagnosis code for rhabdomyolysis, myoglobinuria, and hemoglobinuria (728.88, 791.2, 791.3)or other ICD-9 codes identified during the study
* between the ages of 0-21 years at diagnosis

Exclusion Criteria:

* rhabdomyolysis or serum CK concentrations not actually documented
* patient admitted to the burn center
* patient > 21 years of age

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients diagnosed with rhabdomyolysis/ myoglobinuria/ hemoglobinuria (in-patient, out-patient, ER visit) at a CHMCA facility
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2008-01; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
The presence of rhabdomyolysis based on serum CK concentrations in patients admitted with history of Jimsonweed ingestion. | From admission until discharge

SECONDARY OUTCOMES:
Renal function, liver function, vital signs, physical exam | From admission until discharge

CONTACTS AND LOCATIONS:
Overall Officials: Martha Blackford, Principal Investigator — CHMCA
Locations (1):
- Children's Hospital Medical Center of Akron, Akron, Ohio, United States

REFERENCES:
- [Background] Forrester MB. Jimsonweed (Datura stramonium) exposures in Texas, 1998-2004. J Toxicol Environ Health A. 2006 Oct;69(19):1757-62. doi: 10.1080/15287390600631284. PMID 16905506
- [Background] Ertekin V, Selimoglu MA, Altinkaynak S. A combination of unusual presentations of Datura stramonium intoxication in a child: rhabdomyolysis and fulminant hepatitius. J Emerg Med. 2005 Feb;28(2):227-8. doi: 10.1016/j.jemermed.2004.11.006. No abstract available. PMID 15707824
- [Background] Giannoglou GD, Chatzizisis YS, Misirli G. The syndrome of rhabdomyolysis: Pathophysiology and diagnosis. Eur J Intern Med. 2007 Mar;18(2):90-100. doi: 10.1016/j.ejim.2006.09.020. PMID 17338959